CLINICAL TRIAL: NCT05374616
Title: Natural History Study and Establishment of a Biorepository-TANGO2-related Disorder
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Seema Lalani, Professor, Baylor College of Medicine
Other Study IDs: H-43240
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: TANGO2-related Disorder
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, saliva, skin fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with TANGO2 deficiency: Individuals with TANGO2 deficiency known to have disease causing variants in TANGO2
  Interventions: Genetic: Observation

INTERVENTIONS:
Genetic: Observation — Retrospective and prospective Natural History Study

SUMMARY:
The study aims to establish a biorepository of individuals with TANGO2 deficiency to support scientific research and establish a comprehensive clinical database of affected individuals to understand the disease course.

DETAILED DESCRIPTION:
TANGO2-related disorder is a rare autosomal recessive genetic disorder that can cause recurrent rhabdomyolysis and life-threatening cardiac arrhythmias. Metabolic crises can be triggered by prolonged fasting and dehydration. Intellectual disability, seizures, hypothyroidism, and gait abnormalities are observed frequently. The function of TANGO2 is unknown and the pathogenesis of this disease is poorly understood. Understanding disease mechanism requires studying disease cells/samples and thus establishing a biobank of tissues (blood and fibroblasts) of individuals affected with TANGO2 deficiency is paramount. Natural History Study of TANGO2-related disorder will allow investigators to understand the course of the disease and develop new therapies in the future to decrease morbidity associated with this genetic condition.

ELIGIBILITY:
Inclusion Criteria:

All patients with pathogenic TANGO2 variants will be included.

Exclusion Criteria:

Patients who do not have TANGO2-related disease will be excluded.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with TANGO2-related disorder with any of the following conditions will be recruited: Recurrent rhabdomyolysis, cardiac arrhythmias, muscle weakness, ataxia, progressively unsteady gait, intellectual disability, hypothyroidism, and seizures.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with metabolic and cardiac crisis assessed by the number of hospitalizations | 10 years
  Detailed interview with participants and review of medical records will be used to assess the frequency and triggers of metabolic and cardiac crises

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lalani SR, Liu P, Rosenfeld JA, Watkin LB, Chiang T, Leduc MS, Zhu W, Ding Y, Pan S, Vetrini F, Miyake CY, Shinawi M, Gambin T, Eldomery MK, Akdemir ZH, Emrick L, Wilnai Y, Schelley S, Koenig MK, Memon N, Farach LS, Coe BP, Azamian M, Hernandez P, Zapata G, Jhangiani SN, Muzny DM, Lotze T, Clark G, Wilfong A, Northrup H, Adesina A, Bacino CA, Scaglia F, Bonnen PE, Crosson J, Duis J, Maegawa GH, Coman D, Inwood A, McGill J, Boerwinkle E, Graham B, Beaudet A, Eng CM, Hanchard NA, Xia F, Orange JS, Gibbs RA, Lupski JR, Yang Y. Recurrent Muscle Weakness with Rhabdomyolysis, Metabolic Crises, and Cardiac Arrhythmia Due to Bi-allelic TANGO2 Mutations. Am J Hum Genet. 2016 Feb 4;98(2):347-57. doi: 10.1016/j.ajhg.2015.12.008. Epub 2016 Jan 21. PMID 26805781
- [Background] Miyake CY, Burrage L, Glinton K, Houck K, Hoyos-Martinez A, Graham B, Yang Y, Rawls-Castillo B, Scaglia F, Soler-Alfonso C, Lalani SR. TANGO2 Deficiency. 2018 Jan 25 [updated 2023 Mar 9]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK476443/ PMID 29369572
- [Background] Kremer LS, Distelmaier F, Alhaddad B, Hempel M, Iuso A, Kupper C, Muhlhausen C, Kovacs-Nagy R, Satanovskij R, Graf E, Berutti R, Eckstein G, Durbin R, Sauer S, Hoffmann GF, Strom TM, Santer R, Meitinger T, Klopstock T, Prokisch H, Haack TB. Bi-allelic Truncating Mutations in TANGO2 Cause Infancy-Onset Recurrent Metabolic Crises with Encephalocardiomyopathy. Am J Hum Genet. 2016 Feb 4;98(2):358-62. doi: 10.1016/j.ajhg.2015.12.009. Epub 2016 Jan 21. PMID 26805782
- [Background] Milev MP, Saint-Dic D, Zardoui K, Klopstock T, Law C, Distelmaier F, Sacher M. The phenotype associated with variants in TANGO2 may be explained by a dual role of the protein in ER-to-Golgi transport and at the mitochondria. J Inherit Metab Dis. 2021 Mar;44(2):426-437. doi: 10.1002/jimd.12312. Epub 2020 Sep 21. PMID 32909282
- [Background] Berat CM, Montealegre S, Wiedemann A, Nuzum MLC, Blondel A, Debruge H, Cano A, Chabrol B, Hoebeke C, Polak M, Stoupa A, Feillet F, Torre S, Boddaert N, Bruel H, Barth M, Damaj L, Abi-Warde MT, Afenjar A, Benoist JF, Madrange M, Caccavelli L, Renard P, Hubas A, Nusbaum P, Pontoizeau C, Gobin S, van Endert P, Ottolenghi C, Maltret A, de Lonlay P. Clinical and biological characterization of 20 patients with TANGO2 deficiency indicates novel triggers of metabolic crises and no primary energetic defect. J Inherit Metab Dis. 2021 Mar;44(2):415-425. doi: 10.1002/jimd.12314. Epub 2020 Sep 28. PMID 32929747
- [Background] Powell AR, Ames EG, Knierbein EN, Hannibal MC, Mackenzie SJ. Symptom Prevalence and Genotype-Phenotype Correlations in Patients With TANGO2-Related Metabolic Encephalopathy and Arrhythmias (TRMEA). Pediatr Neurol. 2021 Jun;119:34-39. doi: 10.1016/j.pediatrneurol.2021.02.011. Epub 2021 Mar 8. PMID 33845444
- [Background] Heiman P, Mohsen AW, Karunanidhi A, St Croix C, Watkins S, Koppes E, Haas R, Vockley J, Ghaloul-Gonzalez L. Mitochondrial dysfunction associated with TANGO2 deficiency. Sci Rep. 2022 Feb 23;12(1):3045. doi: 10.1038/s41598-022-07076-9. PMID 35197517